CLINICAL TRIAL: NCT06993961
Title: Ultrasound Measurement of Optic Nerve Sheath Diameter as Non-Invasive Detector of Raised Intracranial Pressure in Adult Traumatic and Non-Traumatic Neurocritical Patients in ICU
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Kareem Elsaeed abdelwahab, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: MD 265/2022
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ultrasound; Optic Nerve Sheath Diameter; Non-Invasive; Intracranial Pressure; Neurocritical; Intensive Care Unit
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patient with suspected high intracranial pressure (ICP) as determined by initial computed tomography (CT) brain.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasound (US) measurement of optic nerve sheath diameter (ONSD) was performed.

SUMMARY:
This study aimed to assess the role of ultrasound as a non-invasive method (bedside) to measure the rise of intracranial pressure by measuring the optic nerve sheath diameter in traumatic and nontraumatic neurocritical patients.

DETAILED DESCRIPTION:
Measurement of intracranial pressure (ICP) is crucial in the management of many neurological conditions. However, due to the invasiveness, high cost, and required expertise of available ICP monitoring techniques, many patients who could benefit from it do not receive it. As a result, a substantial effort has been made to explore and develop novel non-invasive ICP monitoring techniques to improve the overall clinical care of patients suffering from ICP disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Both sexes.
* Patients with suspected high intracranial pressure.

Exclusion Criteria:

* Cases suffering from eye disease or optic nerve problems (Glaucoma, optic Nerve Tumor, Neuritis, Orbital Fracture).
* Patients suffering from mental illness render them incapable of communication & cooperation (For Example: Dementia and irritability).
* Any previous intensive care surgeries & hyperthyroidism (due to exophthalmos)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational prospective trial involved 50 cases aged >18 years old, both sexes, presenting with suspected high intracranial pressure (ICP). The study was conducted from August 2022 to July 2023 after approval from the Ethical Committee of Ain Shams University Hospitals, Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure | 24 hours post-procedure
  Non-invasive bedside intracranial pressure (ICP) assessment via ultrasound (US) measurement of optic nerve sheath diameter (ONSD).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.